CLINICAL TRIAL: NCT06793163
Title: Diagnosis and Allergen Identification of Perioperative Anaphylaxis: a Multicenter Prospective Cohort Study
Brief Title: Diagnosis and Allergen Identification of Perioperative Anaphylaxis
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Chairman of Department of Anesthesiology, Peking University First Hospital
Other Study IDs: 2024-620
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Perioperative/Postoperative Complications; Anaphylaxis; Tryptase; Allergens; Skin Testing
Keywords: Perioperative/Postoperative Complications; Anaphylaxis; Tryptase; Allergens; Skin Testing
MeSH Terms: conditions — Postoperative Complications; Anaphylaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected anaphylaxis: Adult patients with suspected anaphylaxis in the operating rooms, or with history of suspected anaphylaxis in the operating room.

SUMMARY:
Perioperative anaphylaxis may lead to fatal respiratory and/or circulatory events, yet both clinical diagnosis and management are challenging. Serum tryptase is an indicator that can provide important retrospective diagnostic value for anaphylaxis. Another key point in perioperative anaphylaxis management is to identify the allergens, and thus avoid re-exposure during later perioperative management. Skin testing is an important way to identify allergens.

DETAILED DESCRIPTION:
Perioperative anaphylaxis are rare, but may be fatal. The combined use of anesthetic drugs and other medications, and the additional effects of surgical procedures, make the diagnosis and differential diagnosis rather complicated. Subsequent allergy investigations and allergen identification are often difficult.

The change of tryptase levels is an important biomarker in differentiating anaphylaxis from other causes. It is recommended that, in case of any suspicion of perioperative anaphylaxis, serum samples for tryptase detection should be collected as soon as possible after the onset of symptoms and then repeated 24 h later. Skin testing including skin prick tests (SPT) and intradermal tests (IDT) is universally used in identifying allergens. Skin testing will be performed 4-6 weeks after the onset of perioperative anaphylaxis.

This prospective cohort study is designed to clarify the rate of perioperative anaphylaxis with testing serum tryptase level and to identify the underlying allergens by conducting skin testing in surgical patients with suspected perioperative anaphylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2 years or over;
* Suspected anaphylaxis in the operating rooms, or history of suspected anaphylaxis in the operating room.

Exclusion Criteria:

* Refuse to participate;
* Other conditions that are considered unsuitable for study participation.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with suspected anaphylaxis in the operating room.
Sampling Method: Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe perioperative anaphylaxis | On the day of surgery in the operating room
  Perioperative anaphylaxis is defined as anaphylaxis that is confirmed by clinical signs and symptoms and changes of serum tryptase level according to the World Allergy Organization Anaphylaxis Guidance 2020 and occurred in the operating room. Severe perioperative anaphylaxis indicates grade 3 or above according to the World Allergy Organization systemic allergic reaction grading system. The incidence is calculated as the number of cases with severe perioperative anaphylaxis divided by the total number of cases who undergo surgery in the operating room during the study period.

SECONDARY OUTCOMES:
Diagnostic rate of anaphylaxis in patients with suspected perioperative anaphylaxis. | On the day of surgery in the operating room
  Perioperative anaphylaxis is defined as anaphylaxis that is confirmed by clinical signs and symptoms and changes of serum tryptase level according to the World Allergy Organization Anaphylaxis Guidance 2020 and occurred in the operating room.
  The rate is calculated as the number of cases with confirmed anaphylaxis divided by the total number of cases with suspected anaphylaxis in the operating room during the study period.
Incidence of perioperative anaphylaxis | On the day of surgery in the operating room
  Perioperative anaphylaxis is defined as anaphylaxis that is confirmed by clinical signs and symptoms and changes of serum tryptase level according to the World Allergy Organization Anaphylaxis Guidance 2020 and occurred in the operating room. The incidence is calculated as the number of cases with any grade perioperative anaphylaxis divided by the total number of cases who undergo surgery in the operating room during the study period.
Allergen detection in patients with perioperative anaphlaxis | At least 4-6 weeks after the confirmed perioperative anaphylaxis
  Allergen is detected with skin testing in patients with confirmed perioperative anaphylaxis. Skin testing will be performed at least 4-6 weeks after the confirmed anaphylaxis.

OTHER OUTCOMES:
Rate of surgical suspension due to suspected perioperative anaphylaxis. | On the day of surgery suspected perioperative anaphylaxis
  The rate is calculated as the number of patients with surgical suspension due to suspected perioperative anaphylaxis divided by the total number of patients with suspected/confirmed perioperative anaphylaxis in the operating room during the study period.
Rate of unplanned ICU admission due to suspected perioperative anaphylaxis | Within 24 hours of suspected perioperative anaphylaxis
  The rate is calculated as the number of patients with unplanned ICU admission due to suspected perioperative anaphylaxis divided by the total number of patients with suspected/confirmed perioperative anaphylaxis in the operating room during the study period.
Rate of recurrence of perioperative anaphylaxis | On the day of surgery in the operating room
  Perioperative anaphylaxis is defined as anaphylaxis that is confirmed by clinical signs and symptoms and changes of serum tryptase level according to the World Allergy Organization Anaphylaxis Guidance 2020 and occurred in the operating room. The rate is calculated as the number of patients with recurrence of suspected perioperative anaphylaxis divided by the total number of patients with confirmed perioperative anaphylaxis in the operating room during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (4):
- China (4):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Anorectal Hospital (Beijing Erlong Road Hospital）, Beijing, Beijing Municipality
  - Beijing Children's Hospital, Capital Medical University; National Center for Children's Health, China, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Muraro A, Worm M, Alviani C, Cardona V, DunnGalvin A, Garvey LH, Riggioni C, de Silva D, Angier E, Arasi S, Bellou A, Beyer K, Bijlhout D, Bilo MB, Bindslev-Jensen C, Brockow K, Fernandez-Rivas M, Halken S, Jensen B, Khaleva E, Michaelis LJ, Oude Elberink HNG, Regent L, Sanchez A, Vlieg-Boerstra BJ, Roberts G; European Academy of Allergy and Clinical Immunology, Food Allergy, Anaphylaxis Guidelines Group. EAACI guidelines: Anaphylaxis (2021 update). Allergy. 2022 Feb;77(2):357-377. doi: 10.1111/all.15032. Epub 2021 Sep 1. PMID 34343358
- [Background] Tran R, Pedersen K, Kolawole H, Roessler P, Scolaro R. Australian and New Zealand Anaesthetic Allergy Group/Australian and New Zealand College of Anaesthetists perioperative anaphylaxis management guideline 2022. Anaesth Intensive Care. 2024 May;52(3):147-158. doi: 10.1177/0310057X231215823. Epub 2024 Apr 8. PMID 38587791
- [Background] Manian DV, Volcheck GW. Perioperative Anaphylaxis: Evaluation and Management. Clin Rev Allergy Immunol. 2022 Jun;62(3):383-399. doi: 10.1007/s12016-021-08874-1. Epub 2021 Jul 10. PMID 34247332